CLINICAL TRIAL: NCT01273207
Title: Extension Study (Extended Access) of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for the Treatment of Bronchiolitis Obliterans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110064; 11-H-0064
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2019-08-14

CONDITIONS: Bronchiolitis Obliterans; Constructive Bronchiolitis; Graft Versus Host Disease; Bronchiolitis, Exudative; Bronchiolitis, Proliferative; Graft-Versus-Host Disease
Keywords: Peripheral Blood Stem Cell Transplant; Inhaled Cyclosporine; Graft-Versus-Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans; Graft vs Host Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inhaled Cyclosporine in HSCT Participants (Experimental): Hemopoietic Stem Cell transplant (HSCT) subjects with Bronchiolitis Obliterans Syndrome (BOS) received cyclosporine inhalation solution (CIS) at maximum tolerated dose not exceeding 300 mg administered three times per week
  Interventions: Drug: Cyclosporine Inhalation Solution (CIS)

INTERVENTIONS:
Drug: Cyclosporine Inhalation Solution (CIS) — CIS is a sterile, clear, colorless, preservative-free solution of cyclosporine (USP) in propylene glycol developed specifically for administration by oral inhalation.

SUMMARY:
Bronchiolitis Obliterans (BO) is an obstructive lung disease that can affect individuals that have undergone a lung or hematopoietic stem cell transplant. BO has been studied most extensively in lung transplant recipients, where it is considered to represent chronic lung rejection. It is the leading cause of death after lung transplant, with mortality rates up to 55 percent. In hematopoietic stem cell transplantation, BO is thought to be a manifestation of chronic graft-vs-host disease (GVHD). Up to 45 percent of patients undergoing hematopoietic stem cell transplantation at the NHLBI develop a decline in pulmonary function. Conventional therapy for patients who develop BO consists of augmentation of systemic immunosuppressants. Systemic immunosuppression has limited efficacy for BO and is associated with deleterious consequences including increased risk of infections and decreased graft-versus tumor/leukemia effects.

Recently, cyclosporine inhalation solution (CIS) in solution with propylene glycol has been shown to improve overall survival and chronic rejection-free survival in lung transplant patients. These findings suggest targeted delivery of immunosuppressive therapy to the diseased organ warrants further investigation as this may minimize the morbidity associated with systemic immunosuppression. However, there currently exists limited data regarding the overall efficacy of inhaled cyclosporine to treat established BO following lung transplantation. Furthermore, inhaled cyclosporine has not been studied in the treatment of BO following hematopoietic stem cell transplantation.

Here, we propose to evaluate the long-term safety and efficacy, of inhaled CIS for the treatment of BO. Enrollment will be offered to subjects who have completed the end of study (week 18 visit) for the initial protocol (Phase II Trial of CIS in lung transplant and hematopoietic stem cell transplant recipients for treatment of Bronchiolitis Obliterans) and who have shown evidence of benefit (either an improvement or stabilization) in BO/BOS with CIS treatment.

Clinical parameters, including pulmonary function tests, will be measured in addition to laboratory markers of the anti-inflammatory response to CIS. Adverse events associated with extended treatment with CIS will be recorded.

The primary objective is to provide long-term safety and efficacy data for the use of CIS in hematopoietic transplant patients and lung transplant patients with established BO.

Secondary objectives include investigation of the inflammatory pathways that lead to chronic BO and ascertainment of the long term anti-inflammatory effects of this CSA preparation ex vivo and in vivo.

Primary endpoint is the efficacy of extended use CIS for BO/BOS. Secondary endpoints include the toxicity profile (adverse events), improvement in high resolution chest CT images, results of peripheral blood and bronchoalveolar cytokine arrays to assess secondary markers of inflammation, and functional capacity measurements using a six-minute walk test.

DETAILED DESCRIPTION:
Bronchiolitis Obliterans (BO) is an obstructive lung disease that can affect individuals that have undergone a lung or hematopoietic stem cell transplant. BO has been studied most extensively in lung transplant recipients, where it is considered to represent chronic lung rejection. It is the leading cause of death after lung transplant, with mortality rates up to 55 percent. In hematopoietic stem cell transplantation, BO is thought to be a manifestation of chronic graft-vs-host disease (GVHD). Up to 45 percent of patients undergoing hematopoietic stem cell transplantation at the NHLBI develop a decline in pulmonary function. Conventional therapy for patients who develop BO consists of augmentation of systemic immunosuppressants. Systemic immunosuppression has limited efficacy for BO and is associated with deleterious consequences including increased risk of infections and decreased graft-versus tumor/leukemia effects.

Recently, cyclosporine inhalation solution (CIS) in solution with propylene glycol has been shown to improve overall survival and chronic rejection-free survival in lung transplant patients. These findings suggest targeted delivery of immunosuppressive therapy to the diseased organ warrants further investigation as this may minimize the morbidity associated with systemic immunosuppression. However, there currently exists limited data regarding the overall efficacy of inhaled cyclosporine to treat established BO following lung transplantation. Furthermore, inhaled cyclosporine has not been studied in the treatment of BO following hematopoietic stem cell transplantation.

Here, we propose to evaluate the long-term safety and efficacy, of inhaled CIS for the treatment of BO. Enrollment will be offered to subjects who have completed the end of study (week 18 visit) for the initial protocol (Phase II Trial of CIS in lung transplant and hematopoietic stem cell transplant recipients for treatment of Bronchiolitis Obliterans) and who have shown evidence of benefit (either an improvement or stabilization) in BO/BOS with CIS treatment.

Clinical parameters, including pulmonary function tests, will be measured in addition to laboratory markers of the anti-inflammatory response to CIS. Adverse events associated with extended treatment with CIS will be recorded.

The primary objective is to provide long-term safety and efficacy data for the use of CIS in hematopoietic transplant patients and lung transplant patients with established BO.

Secondary objectives include investigation of the inflammatory pathways that lead to chronic BO and ascertainment of the long term anti-inflammatory effects of this CSA preparation ex vivo and in vivo.

Primary endpoint is the efficacy of extended use CIS for BO/BOS. Secondary endpoints include the toxicity profile (adverse events), improvement in high resolution chest CT images, results of peripheral blood and bronchoalveolar cytokine arrays to assess secondary markers of inflammation, and functional capacity measurements using a six-minute walk test.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Completed the End of Study visit (week 19) on the initial protocol (Phase II Trial of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans) in the preceding 12 weeks
  2. Patients have shown evidence for a clinical benefit to CIS as evidenced by one or more of the following:
* Improvement in pulmonary function defined by a 10 percent or more increase in the FEV1 at week 18, confirmed with repeat PFTs at least 1 week apart.
* In patients with progressive disease at study entry on the initial protocol (Phase II Trial of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans), stabilization in pulmonary function, defined as less than a 10 percent improvement in FEV1 or less than 10 percent decline in FEV1 at week 18, confirmed with repeat PFTs at least 1 week apart.
* In patients with stable disease (active BOS stable by FEV1 criteria) at study entry on the initial protocol (Phase II Trial of Cyclosporine Inhalation Solution (CIS) in Lung Transplant and Hematopoietic Stem Cell Transplant Recipients for Treatment of Bronchiolitis Obliterans), stabilization in pulmonary function, defined as less than a 10 percent improvement in their FEV1 or less than 10 percent decline in FEV1, and a decrease in the dose of one or more systemic immunosuppressants by at least 20 percent (sustained for 3 weeks, excluding adjustments made for target drug levels). * The criteria for study entry on this extension protocol are not the same as the criteria for response on the primary protocol to allow for entry of patients on this extension protocol, which is deriving some clinical benefit, but have not met the full response criteria as defined in the primary protocol.

EXCLUSION CRITERIA:

1. More than a 12 week gap in study drug administration (CIS)
2. Evidence of uncontrolled, pulmonary infection
3. ECOG performance status greater than or equal to 3
4. Patient pregnant or breast feeding or not willing to continue the use of an approved method of birth control
5. Life expectancy less than 18 weeks
6. History of hypersensitivity reaction to propylene glycol
7. Documented allergy or intolerance to CIS
8. History of untreated coronary insufficiency, severe cardiac arrhythmias, and/or uncontrolled hypertension.
9. Serum creatinine greater than 2.5 mg/dl
10. Inability to comprehend the investigational nature of the study and provide informed consent

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-03-02 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole J Gormley, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-H-0064.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The lung transplant arm was closed during the study due to lack of subject enrollment
Period: Overall Study
Arm/Group | Inhaled Cyclosporine in HSCT Participants
Started | 7
Completed | 2
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Inhaled Cyclosporine in HSCT Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Status of Pulmonary Disease at Initial Enrollment [Count of Participants; unit: Participants]
  Stable Pulmonary Disease (Stable FEV1) | 4
  Progressive Pulmonary Disease (Declining FEV1) | 3

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Lung Function - Increase in FEV1
Description: Continued improvement in lung function as defined by 10% or more increase in FEV1
Time Frame: 6 Months
Population: Inhaled Cyclosporine in hematopoietic stem cell transplant (HSCT) participants
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Cyclosporine in HSCT Participants
Number analyzed (Participants) | 7
Participants | 0

2. Primary Outcome: Disease Stablization - Decrease in FEV1 or Less Than 10% Increase in FEV1
Description: Stabilization in Pulmonary Function Test (PFT) as defined by less than 10% increase in FEV1 or less than 10% decline in FEV1
Time Frame: 6 Months
Population: Inhaled Cyclosporine in hematopoietic stem cell transplant (HSCT) participants
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Cyclosporine in HSCT Participants
Number analyzed (Participants) | 7
Participants | 7

3. Primary Outcome: Disease Progression - Decrease in FEV1 or Additional/Increase in Immunosuppressive Therapies
Description: Disease progression as defined by a 20% or more decline in FEV1, or those who require an increase in immunosuppressive therapies by at least 25% or the addition of new immunosuppressive therapies.
Time Frame: 6 Months
Population: Inhaled Cyclosporine in hematopoietic stem cell transplant (HSCT) participants
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Cyclosporine in HSCT Participants
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Inhaled Cyclosporine in HSCT Participants
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Cyclosporine in HSCT Participants (N=7)
Post transplant lymphoproliferative disorder (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Body temperature increased (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Sputum culture positive (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Cyclosporine in HSCT Participants (N=7)
Haemoglobinaemia (Blood and lymphatic system disorders) | 2
Oedema peripheral (Cardiac disorders) | 2
Cataract (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Oedema (General disorders) | 1
Influenza (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 2
Breast mass (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dizziness (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT01273207/Prot_SAP_000.pdf